CLINICAL TRIAL: NCT00134888
Title: The Acute and Protracted Blockade Efficacy of Buprenorphine/Naloxone
Brief Title: Blockade Efficacy of Buprenorphine/Naloxone For Opioid Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08045-2; R01-08045-2; DPMC
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2007-07

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
Buprenorphine, a treatment for opioid dependence, can be mixed with naloxone, to limit abuse potential. The purpose of this study is to examine the effectiveness of buprenorphine/naloxone that is given at less than daily intervals, in order to prevent withdrawal symptoms associated with stopping opioid abuse.

DETAILED DESCRIPTION:
Buprenorphine and naloxone are often combined to decrease withdrawal symptoms in opioid dependent individuals. Buprenorphine/naloxone is usually given daily to individuals who are attempting to stop opioid abuse; however, research suggests that individuals may be more inclined to take medication if it is given in less than daily intervals. The purpose of this study is to examine the opioid blockade effects of buprenorphine/naloxone that is administered in less than daily doses to opioid dependent individuals.

This study will last 11 weeks. Participants will stay in a residential research unit for the duration of the study. Participants will be randomly assigned to receive different doses of daily, sublingual buprenorphine/naloxone. After a minimum of 2 weeks on each dose, participants will undergo challenge sessions on each weekday for 1 week (Monday through Friday). Challenge sessions will consist of increasing doses of intramuscular hydromorphone. During the challenge session week, buprenorphine/naloxone will be given only on Monday; a placebo will be given the rest of the week. Challenge sessions will examine the blockade effects of buprenorphine/naloxone at 2, 26, 50, 74, and 98 hours after the last active dose of buprenorphine/naloxone.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for opioid dependence
* Qualifies for opioid substitution treatment (e.g., methadone)

Exclusion Criteria:

* Significant psychiatric or physical disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2000-12; Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Physiological effects | up to one day
drug effects (measured at Week 11) | up to one day

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States